CLINICAL TRIAL: NCT03168581
Title: A Proof of Concept Study to Evaluate Administration of CN-105 in Patients With Acute Supratentorial Intracerebral Hemorrhage
Brief Title: A Proof of Concept Study to Evaluate CN-105 in ICH Patients
Acronym: CATCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AegisCN LLC (Industry)
Collaborators: Duke Clinical Research Institute (Other); PharPoint Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CATCH; 5R01FD005387-02 (FDA)
Record Dates: First submitted 2017-05-02; First posted 2017-05-30 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2019-07

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — apolipoprotein E mimetic peptide CN-105

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CN-105 (Experimental): All eligible subjects will receive study drug, CN-105
  Interventions: Drug: CN-105

INTERVENTIONS:
Drug: CN-105 — Patients with supratentorial intracerebral hemorrhage (ICH) will be evaluated for eligibility within 12 hours of symptom onset. Eligible participants will receive CN-105 administered intravenously (IV) for a 30 -minute infusion every 6 hours for up to a maximum of 3 days (13 doses) or until discharge (if earlier than 3 days)

SUMMARY:
A multicenter, open-label phase 2a trial of CN-105 in patients with supratentorial intracerebral hemorrhage (ICH). Patients will be evaluated for eligibility within 12 hours of symptom onset. Eligible participants (approximately 60) will receive CN-105 administered intravenously (IV) for a 30-minute infusion every 6 hours for up to a maximum of 3 days (13 doses) or until discharge (if earlier than 3 days). Participants will be monitored daily throughout the Treatment phase of the study (up to a maximum of 5 days) and will receive standard-of-care treatment for the duration of the study. Additional protocol assessments will be required during the Treatment phase. After discharge from the hospital, participants will enter a 3-month Follow-up phase, with a clinic visit at 30 days and a follow-up telephone interview with telephone-validated Modified Rankin Scale (mRS) at 90 days after first dose of study agent.

Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent to participate in the study in accordance with required regulations; if a participant is not capable of providing informed consent, written consent must be obtained from the participant's legally authorized representative (LAR).
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Is male or female, age 30 to 80 years, inclusive.
4. Has a confirmed diagnosis of spontaneous supratentorial ICH.
5. Able to receive first dose of study drug ≤ 12 hours after onset of ICH symptoms, such as alteration in level of consciousness, severe headache, nausea, vomiting, seizure, and/or focal neurological deficits, or last-known well time.
6. Has an interpretable and measurable diagnostic CT scan.
7. Has a Glasgow Coma Scale (GCS) score ≥ 5 on presentation
8. Has a National Institutes of Health Stroke Scale (NIHSS) score ≥ 4.
9. Has systolic BP (SBP) < 200 mm Hg at enrollment.

Exclusion Criteria:

1. Is pregnant or lactating.
2. Has a temperature greater than 38.5°C at Screening.
3. Has ICH resulting from trauma.
4. Has infratentorial hemorrhage (any involvement of the midbrain or lower brainstem as demonstrated by radiograph or complete third nerve palsy).
5. Has primary intraventricular hemorrhage deemed to be at high risk for obstructive hydrocephalus, or extra-axial (ie, subarachnoid or subdural) extension of hemorrhage.
6. Has radiographic evidence of underlying tumor.
7. Has an unstable mass or evolving intracerebral compartment syndrome.
8. Has a ruptured aneurysm, arteriovenous malformation, or vascular anomaly.
9. Has a platelet count < 100,000/mL.
10. Has an international normalized ratio (INR) < 1.6 or irreversible coagulopathy either due to medical condition or detected before screening.
11. In the opinion of the investigator is unstable and would benefit from supportive care rather than supportive care plus CN-105.
12. In the opinion of the investigator has any contraindication to the planned study assessments, including CT and MRI.
13. Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which, in the opinion of the investigator, unacceptably increases the individual's risk by participating in the study.
14. Concomitant enrollment in another interventional study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
CN-105 safety assessment | 90 days
  Number and severity of AEs throughout the duration of the study
Mortality | 30 days
  Record In-hospital 30-day mortality
Mortality | 90 days
  record 90-day mortality
In-hospital neurological deterioration | 30 days
  Increase of National Institutes of Health Stroke Scale (NIHSS), > 2 from baseline, persisting more than 24 hours, and unrelated to sedation.

SECONDARY OUTCOMES:
Improvement in 30-day mortality | 30 days
  Compare participants treated with CN-105 with matched controls
Improvement in 30-day functional outcomes | 30 days
  Compare participants treated with CN-105 with matched controls

OTHER OUTCOMES:
Exploratory CT to evaluate progression of edema | 30 days
  To investigate feasibility of noncontrast head computed tomography (CT) as a radiographic surrogate to evaluate progression of perihematomal edema
Exploratory MRI to evaluate progression of edema | 30 days
  To investigate feasibility magnetic resonance imaging (MRI) radiographic surrogate measures to evaluate progression of perihematomal edema
Exploratory neuroinflammatory biomarker assessment to evaluate progression of edema | 90 days
  To investigate feasibility of using serial biochemical markers of neuroinflammation and neuronal injury as a surrogate measure of perihematomal edema and clinical outcome in the setting of spontaneous ICH

CONTACTS AND LOCATIONS:
Overall Officials: Michael L James, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - A.B. Chandler Medical Center-University of Kentucky, Lexington, Kentucky
  - Duke University Health System, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia Health Systems, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guptill JT, Raja SM, Boakye-Agyeman F, Noveck R, Ramey S, Tu TM, Laskowitz DT. Phase 1 Randomized, Double-Blind, Placebo-Controlled Study to Determine the Safety, Tolerability, and Pharmacokinetics of a Single Escalating Dose and Repeated Doses of CN-105 in Healthy Adult Subjects. J Clin Pharmacol. 2017 Jun;57(6):770-776. doi: 10.1002/jcph.853. Epub 2016 Dec 19. PMID 27990643
- [Background] Lei B, James ML, Liu J, Zhou G, Venkatraman TN, Lascola CD, Acheson SK, Dubois LG, Laskowitz DT, Wang H. Neuroprotective pentapeptide CN-105 improves functional and histological outcomes in a murine model of intracerebral hemorrhage. Sci Rep. 2016 Oct 7;6:34834. doi: 10.1038/srep34834. PMID 27713572
- [Derived] Li S, Wangqin R, Meng X, Li H, Wang Y, Wang H, Laskowitz D, Chen X, Wang Y. Tolerability and Pharmacokinetics of Single Escalating and Repeated Doses of CN-105 in Healthy Participants. Clin Ther. 2022 May;44(5):744-754. doi: 10.1016/j.clinthera.2022.03.006. Epub 2022 May 11. PMID 35562205